CLINICAL TRIAL: NCT04349085
Title: Effects of Photobiomodulation Therapy Combined With Static Magnetic Field Applied in Different Moments on Performance and Muscle Recovery in CrossFit® Athletes
Brief Title: Effects of Photobiomodulation Therapy Combined With Static Magnetic Field in CrossFit® Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3.360.743
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Muscle Strength
Keywords: Photobiomodulation Therapy; Low-level Laser Therapy; Static Magnectic Fields; CrossFit®; Strength Training

STUDY DESIGN:
Intervention Model Description: The volunteers will be allocated to four interventions/situation:
  1. Effective PBMT/sMF before WOD and placebo PBMT/sMF after WOD;
  2. Placebo PBMT/sMF before WOD and effective PBMT/sMF after WOD;
  3. Effective PBMT/sMF before WOD and effective PBMT/sMF after WOD;
  4. Placebo PBMT/sMF before WOD and placebo PBMT/sMF after WOD. The order of the interventions will be randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher will program the device (placebo or PMBT) and will be instructed not to inform the volunteers or other researchers as to the type of treatment (PMBT or placebo). Therefore, the researcher responsible for the treatment will be blinded to the type of treatment being administered to the volunteers. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (placebo or PBMT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Effective PBMT/sMF before WOD and Placebo PBMT/sMF after WOD (Experimental): PBMT/sMF will be applied in two steps: effective PBMT/sMF will be applied before the WOD and placebo PBMT/sMF will be applied after the WOD.
  Interventions: Device: Effective PBMT/sMF; Device: Placebo PBMT/sMF
- Placebo PBMT/sMF before WOD and Effective PBMT/sMF after WOD (Experimental): PBMT/sMF will be applied in two steps: placebo PBMT/sMF will be applied before the WOD and effective PBMT/sMF will be applied after the WOD.
  Interventions: Device: Effective PBMT/sMF; Device: Placebo PBMT/sMF
- Effective PBMT/sMF before WOD and Effective PBMT/sMF after WOD (Experimental): PBMT/sMF will be applied in two steps: effective PBMT/sMF will be applied before the WOD and effective PBMT/sMF will be applied after the WOD.
  Interventions: Device: Effective PBMT/sMF
- Placebo PBMT/sMF before WOD and Placebo PBMT/sMF after WOD. (Placebo Comparator): PBMT/sMF will be applied in two steps: placebo PBMT/sMF will be applied before the WOD and placebo PBMT/sMF will be applied after the WOD.
  Interventions: Device: Placebo PBMT/sMF

INTERVENTIONS:
Device: Effective PBMT/sMF — A cluster with 20 diodes, manufactured by Multi Radiance Medical® (Solon, OH, USA), will be used: 4 diodes of 905 nm (1.25 average power, 50 W of peak power for each diode), 8 diodes of 850 nm (40 mW of average power for each diode) and 4 diodes of 633 nm (25 mW average power for each diode). Effective PBMT/sMF will be applied in direct contact with the skin and light pressure in: 4 sites in the knee extensor/hip flexor muscles, 3 sites in the knee flexor/hip extensor muscles and 1 site in the plantar flexor muscles. The effective PBMT/sMF will be applied to both lower limbs. The dose used for applications will be approximately 270 J for knee extensors/hip flexors, 180 J for knee flexors/hip extensors, and 60 J for plantar flexors.
  Arms: Effective PBMT/sMF before WOD and Effective PBMT/sMF after WOD; Effective PBMT/sMF before WOD and Placebo PBMT/sMF after WOD; Placebo PBMT/sMF before WOD and Effective PBMT/sMF after WOD
Device: Placebo PBMT/sMF — A cluster manufactured by Multi Radiance Medical® (Solon, OH, USA) with 20 diodes will be used: Placebo PBMT/sMF will be applied in direct contact with the skin and light pressure in: 4 sites in the knee extensor/hip flexor muscles, 3 sites in the knee flexor/hip extensor muscles and 1 site in the plantar flexor muscles. The placebo PBMT/sMF will be applied to both lower limbs. The dose used for applications will be approximately 0 J per diode. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (active or placebo).
  Arms: Effective PBMT/sMF before WOD and Placebo PBMT/sMF after WOD; Placebo PBMT/sMF before WOD and Effective PBMT/sMF after WOD; Placebo PBMT/sMF before WOD and Placebo PBMT/sMF after WOD.

SUMMARY:
Crossfit® is a method of strength training and fitness built on functional movements, constantly varied and executed at high intensity. Competitions such as the Crossfit® involve physically demanding activities, which in addition to being performed at high intensity also use great measures of aerobic capacity related with performance. These characteristics cause metabolic and muscular stress, as well as a decrease in physical performance. The demand for intensity is the cause of concern regarding the practice of Crossfit® and the risk of injuries. Studies using photobiomodulation therapy combined with static magnetic fields (PBMT/sMF) to delay fatigue and increase performance have obtained positive results in different types of exercise and application times. However, there are no studies investigating the effects of PBMT/sMF in training with similar characteristics as Crossfit®. Therefore, the aim of this project is to verify the effects of PBMT/sMF on performance and muscle recovery of Crossfit® athletes at different times of application (pre workout of the day [WOD] and/or post WOD) in order to determine the best way to use the therapy.

DETAILED DESCRIPTION:
To achieve the proposed objective it will be performed a randomized, crossover, triple-blind (volunteers, outcome assessors and therapists), placebo-controlled trial.

Twelve volunteers will be allocated to four interventions/situation. The order of the interventions/situations will be randomized.

The volunteers will be treated by a blinded therapist.

The outcomes will be obtained at baseline (prior to WOD), and 1 hour, 24 and 48 hours after WOD. Except for the ratings of perceived exertion that will be obtained at baseline, after WOD, and 1 hour, 24 and 48 hours after WOD. In addition, for the functional analysis the data will be collected at baseline, after applied intervention, and 1 hour, 24 and 48 hours after WOD. The data will be collected by a blinded assessor.

The WOD will be consisted in finish as quickly as possible a sequence of three exercises (Calories in Assault AirBike®, Hang Squat Clean and Box Jump Over), in a well-known series model for the athletes, without rest.

The investigators will analyze: ratings of perceived exertion; activity of creatine kinase (CK); levels of the cytokine Interleukin-6 (IL-6), and maximum number of free squat reps in 1 minute.

Statistical analysis:

All data will be analyzed both in their absolute values and in relation to their percentage variation from the values obtained in the pre-WOD (baseline) assessments. The results obtained will be tested for normality using the Kolmogorov-Smirnov test. If data show normal distribution, the ANOVA test (one or two way depending on the outcome analyzed) with post-hoc Bonferroni will be used. The level of statistical significance will be p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Crossfit® amateur male athletes;
* who did not present a history of musculoskeletal injury in the regions of the hips, knees and calves in the month preceding the study;
* who were not using pharmacological agents;
* athletes should have been practicing the sport for at least 1 year;
* voluntarily commit to participate in all stages.

Exclusion Criteria:

* who presented musculoskeletal or joint injuries during data collection.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Change in functional capacity | 1 minute post-treatment, 1hour, 24 hours and 48 hours after WOD (workout of the day).
  The functional capacity will be measured by a maximum number of free squat repetitions within 1 minute.

SECONDARY OUTCOMES:
Perception of exercise intensity | 1 minute after WOD, 1 minute post-treatment, 1 hour, 24 hours and 48 hours after WOD (workout of the day).
  The perception of exercise intensity will be measured by a 0-100 Ratings of Perceived Exertion Scale: in this scale lower score, means lower degree of fatigue and higher score, means higher degree of fatigue.
Activity of creatine kinase (CK) | 1 hour, 24 hours and 48 hours after WOD (workout of the day).
  The activity of CK will be analyzed by spectrophotometry and using specific reagent kits from the blood samples collected.
Levels of interleukin-6 (IL-6) | 1 hour, 24 hours and 48 hours after WOD (workout of the day).
  The levels of interleukin-6 will be analyzed by enzyme-linked immunosorbent assay (ELISA) and using specific reagent kits from the blood samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar Pinto Leal Junior, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request addressed to the principal investigator
Supporting Information: Study Protocol, SAP, CSR